CLINICAL TRIAL: NCT06175429
Title: Prognostic Value of Exhaled Isoprene Levels for Morbidity and Functional Outcome in Cardiosurgical Patients - A Single Center Prospective Observational Cohort Study
Brief Title: Prognostic Value of Exhaled Isoprene Levels for Morbidity and Functional Outcome in Cardiosurgical Patients
Acronym: PREDICT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Rostock (Other)
Collaborators: Prof. Dr. Daniel A. Reuter, Head of Department, Department of Anesthesiology, Intensive Care Medicine and Pain Therapy, Rostock University Medical Center (Unknown); Prof. Dr. Christian D. Etz, Head of Department, Department of Cardiac Surgery, Rostock University Medical Center (Unknown); PD Dr. Johannes Ehler, Consultant, Department of Anesthesiology and Intensive Care Medicine, University Hospital Jena (Unknown)
Responsible Party: Principal Investigator, Felix Klawitter, MD, Dr. med. Felix Klawitter, DESAIC, University of Rostock
Other Study IDs: PREDICT
Record Dates: First submitted 2023-11-29; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Frailty; Muscle Weakness; Volatile Organic Compounds; Isoprene
MeSH Terms: conditions — Frailty; Muscle Weakness | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac surgery: Patients undergoing elective cardiac surgery
  Interventions: Diagnostic Test: Physical performance testing; Diagnostic Test: Breath sampling and VOC analysis; Diagnostic Test: Muscle ultrasound; Diagnostic Test: Blood-based biomarker analysis

INTERVENTIONS:
Diagnostic Test: Physical performance testing — Assessment of physical performance using established clinical tests and scoring systems
Diagnostic Test: Breath sampling and VOC analysis — Sampling of exhaled breath and using Proton-transfer-reaction time-of-flight mass spectrometry (PTR-TOF) for VOC quantification.
Diagnostic Test: Muscle ultrasound — Quantitative and qualitative assessment of different limb skeletal muscles using non-invasive ultrasound.
Diagnostic Test: Blood-based biomarker analysis — Blood sampling and assessment of different blood-based biomarkers of muscle integrity using Enzyme-linked Immunosorbent Assay (ELISA) and Electrochemiluminescence Immunoassay (ECLIA)

SUMMARY:
The perioperative preservation of functionality and quality of life plays an increasingly important role in older physically limited and frail patients undergoing cardiac surgery. Hereby, impairments of the skeletal muscle system integrity often contributes to a reduced physical performance. Early identification of these high-risk patients could help to initiate appropriate preventive and therapeutic measures. Volatile organic compounds (VOC) represent a non-invasive and real-time measurable approach for recording physiological and pathophysiological processes. Isoprene (2-methyl-1,3-butadiene) is one of the most abundantly exhaled VOCs and has recently been shown to originate from skeletal muscle metabolism. However, the prognostic value of isoprene as a volatile biomarker for skeletal muscle integrity, physical performance and functional outcome in patients undergoing cardiac surgery has not been evaluated before.

DETAILED DESCRIPTION:
This is a single center prospective observational study evaluating exhaled isoprene as a perioperative volatile biomarker of skeletal muscle integrity, physical performance and functional outcome in cardiosurgical patients. All study participants will be assessed by comprehensive clinical examinations, laboratory testing, breath analysis and skeletal muscle ultrasound before, during as well as five and thirty days after surgery. Clinical assessments will be performed using established clinical scores and scales (e.g. the Short Physical Performance Battery and the Fried Frailty Index). Laboratory testing comprises a broad panel of blood-based biomarkers of skeletal muscle integrity and metabolism.

The investigators hypothesize that:

* perioperative exhaled isoprene levels correlate with postoperative measures of physical performance, functional outcome and morbidity
* perioperative exhaled isoprene levels differ between patients with and without physical frailty
* perioperative exhaled isoprene levels correlate with sonographic and laboratory parameters of skeletal muscle integrity

ELIGIBILITY:
Inclusion Criteria:

* Age >= 65 years
* planned cardiac surgery
* operation duration >60 min

Exclusion Criteria:

* refusal of study participation
* emergency / urgent surgery
* acute myocardial infarction
* acute or chronic infection
* Pre-existing illness with permanent restriction of mobility
* Pre-existing neuromuscular disease
* current malignant disease
* terminal renal insufficiency
* severe liver cirrhosis
* severe obstructive pulmonary disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients undergoing elective cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery | day 5 after surgery
  Assessment of patient's physical performance using the Short Physical Performance Battery (SPPB, Score, scales 0-12), whereby a higher SPPB corresponds to a better physical performance.

SECONDARY OUTCOMES:
Cumulated Ambulation Score | days 5 and 30 after surgery
  Assessment of functional patient outcome using the Cumulated Ambulation Score (CAS, Score, scales 0-6), whereby a higher CAS corresponds to a better functional outcome.
Morbidity | day 30 after surgery
  Assessment of the cumulative number of postoperative complications after surgery.
Isoprene concentration in patients with and without frailty | day 5 after surgery
  Comparison of exhaled isoprene levels (concentrations, part per billion volume - ppbV) measured by PTR-TOF between patients with and without physical frailty.
Medical Research Council Sum Score | day 5 after surgery
  Assessment of general muscle strength of study participants using the Medical Research Council Sum Score (MRCSS, Score, scales 0-60), whereby a higher MRCSS corresponds to a higher muscle strength.
Muscle thickness | day 5 after surgery
  Assessment of muscle thickness (mm) using muscle ultrasound in eight different limb skeletal muscles.
Concentrations of blood-based biomarkers | day 5 after surgery
  Assessment of blood-based biomarker concentrations (pmol/l) of skeletal muscle integrity and metabolism.

CONTACTS AND LOCATIONS:
Overall Officials: Felix Klawitter, Dr. med., Principal Investigator — Department of Anesthesiology, Intensive Care Medicine and Pain Therapy, Rostock University Medical Center
Locations (1):
- Department of Anesthesiology, Intensive Care Medicine and Pain Therapy, Rostock University Medical Center, Rostock, Mecklenburg-Vorpommern, Germany